CLINICAL TRIAL: NCT03396991
Title: Comparative Evaluation of Two Different Post-Operative Analgesia After Hallux Valgus Correction in One-day Surgery Patients
Brief Title: Comparative Evaluation of Two Different Post-Operative Analgesia After Hallux Valgus Correction
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FERRONE GIULIANO, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 50990/17
Record Dates: First submitted 2017-12-29; First posted 2018-01-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
Keywords: Analgesia technique; Pain control
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: In the study Group the investigators enrolled 26 patients scheduled for hallux valgus surgery and treated with a new analgesici approach. After sub-gluteal sciatic nerve block with short acting local anesthetic (mepivacaine 2%, 15 ml), each patient received an ultrasound-guided Posterior Tibial Nerve Block (PTNB) with levobupivacaine 0,5% (7-8 ml). The investigators measured: the intensity of pain at the baseline (before the surgery) and at 3, 6, 12 and 24 hours (h) using a Visual Analogue Scale (VAS); the consumption of oxycodone in the first 24 hours after surgical treatment and the motor recovery using modified Bromage score.
- Control group: The investigators compared the study group with a control group of 26 patients previously scheduled for the same surgery and treated with another post-operative analgesia technique more frequently used in our hospital: local infiltration (Local Infiltration Anesthesia, LIA) with levobupivacaine 0, 5% (15 ml) performed by the surgeon directly on the operative site.

SUMMARY:
Background: Recent studies showed the efficiency of several techniques of anesthesia in foot surgery. The new mini-invasive surgical approaches should require less analgesia and rapid motor recovery after surgery. The aim of this study was the evaluation of two different techniques on postoperative analgesia and motor recovery after hallux valgus correction in one-day surgery patients.

DETAILED DESCRIPTION:
The hallux valgus surgery is often characterized by a significant post-operative pain difficult to control with oral analgesics. Consequently, large doses of parenteral opioids are often required Various nerve blocks (popliteal, saphenous, sciatic) can give excellent post-operative pain control. Among loco-regional anesthesia techniques, the sciatic nerve block provides good post-operative pain relief after foot surgery. Thus, sciatic nerve block with long-acting local anesthetics (with or without a peri-neural catheter) has been recommended as a primary option. This analgesic approach should cause a difficult discharge in ambulatory and one-day surgery patients, due to the prolonged motor recovery and loss of proprioception and protective pain reflexes. Therefore, it would be preferable to use the sciatic nerve block just for intra- operative anesthesia without affecting motor recovery, and to apply multimodal analgesia for post- operative pain management. Hallux valgus repair can now be done percutaneously, a minimally invasive technique called ''mini-invasive hallux valgus repair'', consisting in osteotomies through 3 to 5 mm incisions, without internal fixation. This approach requires less dissection and exposure, determining a smaller inflammatory response and theoretically causing less pain. Ideal anesthesia for these procedures should provide rapid patient recovery, minimal nursing care requirements in the post- anesthesia care unit and an earlier hospital discharge. It must provide effective analgesia, since the foot surgery is known to induce a moderate-to- severe post-operative pain, that represents one of the major limitations to hospital discharge on the day of surgery and is the main cause of re-admission.

The aim of this matched-control study was to evaluate two different techniques of post-operative analgesia after hallux valgus correction in one-day surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* hallux valgus deformity
* pain
* walking difficulty with shoes

Exclusion Criteria:

* peripheral circulatory disorders
* foot skin lesion
* local anesthetic allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: twenty-six consecutive ASA physical status I or II ambulatory patients (study group, SG) scheduled for elective hallux valgus surgery were enrolled. All patients had unilateral procedures
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Pain control measured by a visual analogue scale of Scott-Huskisson (VAS score) | One month
  Pain control measured by a visual analogue scale of Scott-Huskisson (VAS, 0 lack of pain, 10 the worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Ferrone, Principal Investigator — Fondazione policlinico Gemelli
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singelyn FJ. Single-injection applications for foot and ankle surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):247-54. doi: 10.1053/bean.2002.0236. PMID 12491555
- [Background] Turan I, Assareh H, Rolf C, Jakobsson J. Multi-modal-analgesia for pain management after Hallux Valgus surgery: a prospective randomised study on the effect of ankle block. J Orthop Surg Res. 2007 Dec 18;2:26. doi: 10.1186/1749-799X-2-26. PMID 18088436
- [Background] Samuel R, Sloan A, Patel K, Aglan M, Zubairy A. The efficacy of combined popliteal and ankle blocks in forefoot surgery. J Bone Joint Surg Am. 2008 Jul;90(7):1443-6. doi: 10.2106/JBJS.G.01133. PMID 18594091